CLINICAL TRIAL: NCT05207995
Title: A Phase ½ Study to Evaluate the Safety and Feasibility of Autologous Tolerogenic Dendritic Cells in Patients With Type 1 Diabetes Mellitus
Brief Title: The Treatment of Patients With Type 1 Diabetes Mellitus With Autologous Tolerogenic Dendritic Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: Belarusian State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_DM
Record Dates: First submitted 2021-11-29; First posted 2022-01-26 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Type 1 Diabetes Mellitus receiving standard treatment and Tolerogenic Dendritic Cells (Experimental): Group 1: Patients with Type 1 Diabetes Mellitus receiving standard treatment and Tolerogenic Dendritic Cells
  Interventions: Biological: Autologous tolerogenic dendritic cells; Other: Standard treatment according to the clinical protocols
- Patients with Type 1 Diabetes Mellitus receiving standard treatment (Active Comparator): Group 2: Patients with Type 1 Diabetes Mellitus receiving standard treatment
  Interventions: Other: Standard treatment according to the clinical protocols

INTERVENTIONS:
Biological: Autologous tolerogenic dendritic cells — Autologous tolerogenic dendritic cells treated with Vitamin-D3, co-cultivated with mesenchymal stem cell and primed peptides (MSC-tolDC) injected subcutaneous.
  Arms: Patients with Type 1 Diabetes Mellitus receiving standard treatment and Tolerogenic Dendritic Cells
Other: Standard treatment according to the clinical protocols — Standard treatment of type 1 diabetes mellitus according to the clinical protocols

SUMMARY:
The purpose of this study is to determine the safety and tolerability of the administration of tolerogenic dendritic cells in patients with type 1 diabetes mellitus.

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety and tolerability of the administration of autologous monocyte-derived dendritic cells tolerised with Vitamin-D3, co-cultivated with mesenchymal stem cell and primed peptides in patients with type 1 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 1 Diabetes Mellitus
* The patient can read, understand, follow the examination procedures and complete, if necessary, the required documentation
* Written informed consent

Exclusion Criteria:

* The presence of any malignant tumor within the last 5 years
* Acute or chronic diseases in the stage of decompensation
* Chronic infectious diseases: HIV, viral hepatitis B, C, tuberculosis
* Patients who are pregnant, breastfeeding, or fertile patients who are not using adequate contraceptive methods
* Chronic and protracted mental disorders, all diseases with the presence of the syndrome of dependence on alcohol, drugs and psychoactive substances, any other condition that makes the patient unable to understand the nature, extent and possible consequences of the study or, in the opinion of the researcher, prevents the patient from observing and performing protocol
* Patients are unable or unwilling to give written informed consent and / or follow research procedures
* Any other medical condition that, in the opinion of the investigator, may be associated with an increased risk to the patient or may affect the outcome or evaluation of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
The glucose concentration in blood | 1 month
  To assess the glucose concentration in blood
The glycated hemoglobin concentration | 1 month
  To assess the β-cell function measured by the glycated hemoglobin in blood
The C-peptide level in blood | 1 month
  To assess the β-cell function measured by the C-peptide level
The glucose concentration in blood | 6 months
  To assess the glucose concentration in blood
The glycated hemoglobin concentration | 6 months
  To assess the β-cell function measured by the glycated hemoglobin in blood
The C-peptide level in blood | 6 months
  To assess the β-cell function measured by the C-peptide level
The glucose concentration in blood | 1 year
  To assess the glucose concentration in blood
The glycated hemoglobin concentration | 1 year
  To assess the β-cell function measured by the glycated hemoglobin in blood
The C-peptide level in blood | 1 year
  To assess the β-cell function measured by the C-peptide level
Autoantigen specific T cell count | 1 month
  To determine the autoantigen specific T cell count using the flow cytometry
Autoantigen specific T cell count | 6 months
  To determine the autoantigen specific T cell count using the flow cytometry
Autoantigen specific T cell count | 1 year
  To determine the autoantigen specific T cell count using the flow cytometry
Adverse effects associated with the therapy | 1 month
  Determination of adverse effects associated with the therapy
Adverse effects associated with the therapy | 1 year
  Determination of adverse effects associated with the therapy

CONTACTS AND LOCATIONS:
Overall Officials: antonevich.n@gmail.com Antonevich, Dr, Study Director — the Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus; Tatiana Mokhort, Prof, Study Director — Belarusian State Medical University; Andrei Y Hancharou, Dr., Study Director — The Institute for Biophysics and Cell Engineering of the NAS of Belarus; Yana S Minich, Principal Investigator — The Institute for Biophysics and Cell Engineering of the NAS of Belarus
Locations (1):
- Healthcare institution "Minsk City Clinical Endocrinology Center", Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No